CLINICAL TRIAL: NCT06427772
Title: Incidence of Early Infection After Bipolar Hemiarthroplasty and Its Associated Factors in Fracture Neck of Femur
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Sallam Abo El-azaiem Mohamed, principal investigator, Assiut University
Other Study IDs: Sallam
Record Dates: First submitted 2024-05-15; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Prosthetic-joint Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1 diseased group(infected): the presence of persistent discharge after 7 days diagnostic for early infection follow up period first 4 week postoperative bipolar hemiarthroplasty in fracture neck of femur study the risk factors in this group
  Interventions: Procedure: bipolar hemiarthroplasty
- group 2 : control group (normal ): no infection after hemiarthroplasty follow up period first 4 week postoperative bipolar hemiarthroplasty in fracture neck of femur
  Interventions: Procedure: bipolar hemiarthroplasty

INTERVENTIONS:
Procedure: bipolar hemiarthroplasty — bipolar hemiarthroplasty for neck femur fracture

SUMMARY:
Periprosthetic joint infections (PJI) following hemiarthroplasty for hip fractures are a catastrophic complication that results in severe worsening of patients' daily function and quality of life. The incidence of prosthetic joint infection (PJI) in hemiarthroplasty after femoral neck fracture varies from 2% to 17%. Identifying risk factors associated with early infection following HA for hip fractures may provide an opportunity to treat and prevent this potential complication with preoperative planning in many patients. So investigators will study the rate of early infection and its associated factor after bipolar hemiarthroplasty.

DETAILED DESCRIPTION:
Femoral neck fractures (FNF) have a significant incidence and a rising trend worldwide. FNF is associated with a high mortality and disability rate, decreasing the independence and quality of life for affected patients. Acute displaced intracapsular femoral neck fractures account for about half of all hip fractures, with the majority of these fractures in older patients being treated surgically with hip hemiarthroplasty(HA), total hip arthroplasty, or internal fixation. Hemiarthroplasty is also used to treat femoral neck nonunion, failed screw fixation, and pathological femoral neck fracture. The treatment aims are to reduce pain, allow early mobilization, and restore the patient's pre-injury level of function while limiting perioperative surgical and medical complications. Patients with FNF frequently undergo hemiarthroplasty to restore joint biomechanics. Two types of implants are used in hemiarthroplasty: monopolar and bipolar . The bipolar implants have a polyethylene bearing between the stem and head of the endoprosthesis, which allows the components to rotate. There are debatable findings and a lack of consensus on the optimal component for hemiarthroplasty. Periprosthetic joint infections (PJI) following hemiarthroplasty for hip fractures are a catastrophic complication that results in severe worsening of patients' daily function and quality of life. The incidence of prosthetic joint infection (PJI) in hemiarthroplasty after femoral neck fracture varies from 2% to 17%. Identifying risk factors associated with early infection following HA for hip fractures may provide an opportunity to treat and prevent this potential complication with preoperative planning in many patients. So investigators will study the rate of early infection and its associated factor after bipolar hemiarthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients with femoral neck fractures and treated by bipolar hemiarthroplasty.
* Patients or their legal representative able to give informed consent.

Exclusion Criteria:

* Patients that received HA secondary to a failed internal fixation of a femoral neck fracture.
* Patients with a pathological fracture due to malignancy.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: * Study Setting: Department of Orthopedic and Trauma Surgery, Assiut University.
  * Study subjects:
    a. Inclusion criteria:
  * Patients with femoral neck fractures and treated by bipolar hemiarthroplasty.
  * Patients or their legal representative able to give informed consent. b. Exclusion criteria:
  * Patients that received HA secondary to a failed internal fixation of a femoral neck fracture.
  * Patients with a pathological fracture due to malignancy.
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
incidence of early infection after bipolar hemiarthroplasty | 4 weeks postoperative
  investigators will take all cases with bipolar hemiarthroplasty after femoral neck fracture then follow up them for 4 weeks. An infection was categorized as early, if it occurred within 4 weeks after surgery After that investigators will classify them to infected (disease group) and non infected (control group) and studying risk factor predisposing to early infection after HA.
  For diagnosis of infection : the presence of persistent discharge after 7 days
risk factor predisposing to early infection after HA.1-preoperative parameters :Patient age | preoperative evaluation 1 week
  Age in years
risk factor predisposing to early infection after HA.1-preoperative parameters :sex | preoperative evaluation 1 week
  male or female
risk factor predisposing to early infection after HA.1-preoperative parameters :Chronic diseases as Diabetes, rheumatoid arthritis and other inflammatory or autoimmune arthritis. | preoperative evaluation 1 week
  present or not
risk factor predisposing to early infection after HA.1-preoperative parameters : • Active skin disease (at site of surgical incision) | preoperative evaluation 1 week
  present or not
risk factor predisposing to early infection after HA.1-preoperative parameters : • Smoking and alcohol consumption | preoperative evaluation 1 week
  yes or no
risk factor predisposing to early infection after HA.1-preoperative parameters : • Distant septic focus after arthroplasty as (pneumonia ,UTI ,abdominal ,oral and cutaneous infection). | preoperative evaluation 1 week
  present or no
risk factor predisposing to early infection after HA.2-intraoperative parameters : • Surgery time . | at time of operation
  in hours
risk factor predisposing to early infection after HA.2-intraoperative parameters :• Appropriate antibiotics prophalyxis and Need to blood transfusion. | at time of operation
  yes or no
risk factor predisposing to early infection after HA.3-postoperative parameters :• Persistent drainage after 7 days. | 1 week postoperative
  time in days